CLINICAL TRIAL: NCT01513278
Title: Randomized, Double-blind, Split-body, Placebo-controlled Phase Ib Study of APN201 (Liposomal Recombinant Human Cu/Zn-superoxide Dismutase) for the Prevention of Radiation-induced Dermatitis in Women With Breast Cancer
Brief Title: Study of APN201 (Liposomal Recombinant Human Cu/Zn-Superoxide Dismutase) for the Prevention of Radiation-induced Dermatitis in Women With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apeiron Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APN201-1-01
Record Dates: First submitted 2011-12-14; First posted 2012-01-20 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Radiation Induced Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Placebo Comparator): All patients receive APN201 and placebo at the same time. The irradiated region is divided vertically into two symmetric areas (left and right). One area is treated with APN201, the other area is treated with placebo (empty liposomes formulated as a hydrophilic gel) in a double-blind fashion.
  Interventions: Drug: APN201; Drug: Placebo
- APN201 (Active Comparator): APN201 (recombinant human superoxide dismutase (rhSOD) encapsulated in liposomal vesicles formulated as a hydrophilic gel)
  Interventions: Drug: APN201

INTERVENTIONS:
Drug: APN201 — All patients receive APN201 and placebo at the same time. The irradiated region is divided vertically into two symmetric areas (left and right). One area is treated with APN201 (recombinant human superoxide dismutase (rhSOD) encapsulated in liposomal vesicles formulated as a hydrophilic gel; 1.6 mg rhSOD per mL), the other area is treated with placebo (empty liposomes formulated as a hydrophilic gel) in a double-blind fashion.
  Study treatment (APN201 and placebo) starts on the day of initiation of radiation therapy and continues until the end of radiation therapy to the whole breast (25 or 28 daily fractions to a total dose of 50.0 Gy or 50.4 Gy, respectively). Study treatment is applied as a thin film on the irradiated area ≥10 minutes each day before radiation therapy (approximately 1 mL APN201 per 100 cm2 of the radiation field size and approximately 1 ml placebo per 100 cm2 of the radiation field size).
Drug: Placebo — All patients receive APN201 and placebo at the same time. The irradiated region is divided vertically into two symmetric areas (left and right). One area is treated with APN201 (recombinant human superoxide dismutase (rhSOD) encapsulated in liposomal vesicles formulated as a hydrophilic gel; 1.6 mg rhSOD per mL), the other area is treated with placebo (empty liposomes formulated as a hydrophilic gel) in a double-blind fashion.
  Study treatment (APN201 and placebo) starts on the day of initiation of radiation therapy and continues until the end of radiation therapy to the whole breast (25 or 28 daily fractions to a total dose of 50.0 Gy or 50.4 Gy, respectively). Study treatment is applied as a thin film on the irradiated area ≥10 minutes each day before radiation therapy (approximately 1 mL APN201 per 100 cm2 of the radiation field size and approximately 1 ml placebo per 100 cm2 of the radiation field size).
  Arms: Control arm

SUMMARY:
The standard treatment for early-stage breast cancer is breast-conserving surgery followed by adjuvant radiation therapy to the whole breast. This approach leads to low recurrence rates with a good cosmesis and provides an effective alternative to mastectomy. However, in most women receiving radiotherapy radiation dermatitis occur to some degree.

Radiation dermatitis generally manifests within a few weeks after the start of radiation therapy. Its onset varies depending on the radiation dose intensity and the normal tissue sensitivity of individuals. As the cumulative dose of radiation increases the transient erythema occurring during the first weeks of radiotherapy may evolve into the more persistent erythema and to dry or even moist desquamation that reflects the damage to the basal cell layer and the sweat and sebaceous glands.

There is currently no evidence that prophylactic treatments, beyond keeping the irradiated area clean and dry, are effective in reducing the incidence or severity of radiation dermatitis (Bolderston et al. 2006).

However, together with other enzymes of the peroxidase pathway, SOD scavenges the superoxide, hydroxyl, and other oxygenated free radicals (Klug et al. 1972; Tainer at al. 1983). In physiological conditions, the production of free radicals (Monte & Sacerdote 1994) and the action of antiradicals' enzymes is balanced. Following tissue injuries, either pathological or caused by agents such as radiation therapy, an excess production of free radicals is observed (Petkau 1986; Lorette & Machet 2001). Furthermore, basal SOD is increased in breast cancer patients before radiation therapy as compared to controls (Seth et al. 2003), and decreases after radiotherapy (Ray at al. 2000). Hence, liposomal rhSOD applied during radiotherapy could be used to prevent the effects of free radicals and thus might protect the patient's skin from radiation-induced skin reactions.

TREATMENT PLAN All patients receive APN201 and placebo at the same time. The irradiated region is divided vertically into two symmetric areas (left and right). One area is treated with APN201, the other area is treated with placebo in a double-blind fashion.

Study treatment (APN201 and placebo) starts on the day of initiation of radiation therapy and continues until the end of radiation therapy to the whole breast (25 or 28 daily fractions to a total dose of 50.0 Gy or 50.4 Gy, respectively) (see schedule of assessments, section 5.1).

Study treatment is stopped if radiation dermatitis of ≥ grade 2 occurs in one or both treated areas for ≥ 3 days AND a difference in the severity of radiation dermatitis of ≥ 1 grade is seen between the two treated areas. From that point in time the patient only receives the treatment that appeared to be beneficial and this treatment is applied to the whole irradiated region until completion of the 25th, respectively 28th, fraction.

Treatment stops earlier in case of progressive disease or unacceptable toxicity or intolerability.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age, with breast cancer, treated by breast conserving surgery and scheduled to receive adjuvant radiotherapy to the breast alone
* Bra cup size ≤D
* Karnofsky performance status of ≥ 80%
* Women of childbearing potential must have a negative pregnancy test before study entry and must agree to use a medically acceptable method of birth control throughout the study period
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Bilateral breast cancer
* Inflammatory breast cancer
* Lymphangiosis carcinomatosa
* Medically significant dermatologic conditions affecting the irradiated area
* Planned use of other agents with the aim of preventing and/or treating radiation dermatitis
* Concomitant medications which might exacerbate radiation dermatitis
* History of previous radiation therapy of the breast
* Pregnancy or breastfeeding
* Having received any other investigational agent within 4 weeks before enrolment
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of APN201 | From baseline until 1 day following the final radiotherapy fraction, assessed for a maximum of 28 radiotherapy fractions.
  Adverse events, vital signs and laboratory assessments (hematology, serum chemistry) are used for safety evaluations.

SECONDARY OUTCOMES:
To evaluate the efficacy of APN201 in the prevention of radiation-induced dermatitis | From baseline until 1 day after the final radiotherapy fraction, assessed for a maximum of 28 radiotherapy fractions.
  The following parameters are used for efficacy evaluations:
  * Time to ≥ grade 2 radiation dermatitis
  * Incidence of ≥ grade 2 radiation dermatitis
  * Severity of radiation dermatitis
  * Pain intensity (pain on touching the skin) due to radiation therapy
  * Irradiated skin evaluations using the digital wound documentation system W.H.A.T. (wound healing analysing tool) and a spectrophotometer

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz; Department of Therapeutic Radiology and Oncology, Graz, Austria, Austria